CLINICAL TRIAL: NCT05514548
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of the Efficacy, Safety, and Pharmacokinetics of Two Doses of INV-202 in Patients With Diabetic Kidney Disease
Brief Title: Phase 2 Study of INV-202 in Patients With Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inversago Pharma Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INV-CL-106
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Type 1 diabetes mellitus (T1DM); Type 2 diabetes mellitus (T2DM)
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- INV 202 10 mg (Experimental): INV-202 10 mg Arm
  Interventions: Drug: INV-202
- INV-202 25 mg (Experimental): INV-202 25 mg Arm
  Interventions: Drug: INV-202
- Placebo (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INV-202 — INV-202 is a new generation of CB1R antagonist developed by Inversago for potential use as a therapeutic method for the treatment of metabolic disorders, including nonalcoholic steatohepatitis, diabetes and its complications (such as DKD), and hypertriglyceridemia.
  Other Names: None applicable
  Arms: INV 202 10 mg; INV-202 25 mg
Drug: Placebo — Placebo Matching size and number of tablets
  Other Names: None applicable
  Arms: Placebo

SUMMARY:
The study is designed to assess the efficacy, safety, tolerability, and transformation within the human body of INV-202 investigational drug in the treatment of adult participants with a diagnosis of Diabetic Kidney Disease due to either Type 1 diabetes mellitus or Type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo controlled, dose ranging, multicenter study designed to assess the efficacy, safety, tolerability, and pharmacokinetics of INV-202 for the treatment of adult participants with a diagnosis of DKD due to either Type 1 diabetes mellitus (T1DM) or Type 2 diabetes mellitus (T2DM) (diagnosed ≥1 year) who are on a stable anti diabetic medication regimen for ≥4 months prior with a HbA1c <9.5%. Approximately 240 participants (80/arm) will be randomized to 1 of 3 treatment arms in a 1:1:1 ratio: INV 202 10 mg, INV-202 25 mg, or placebo. The assigned study treatment will be taken once daily (QD), for 16 weeks.

Due to the high expected screen failure rates, participants may be pre-screened at sites with an approved pre-screening ICF.

Each participant will be allowed 1 retest during the screening period if they fail screening and 1 re-screening on a case by case basis with approval from the Worldwide medical monitors.

Study participation will last approximately 22 weeks and includes a Screening Period (up to 4 weeks), a Study Treatment Period with 16 weeks of daily study treatment, and a Safety Follow-Up Visit consisting of a phone call 2 weeks after the End of Treatment Visit (Week [W]18) to allow reporting of any adverse events following withdrawal of the study drug.

Any participant who withdraws before completing treatment will be requested to return for an Early Termination Visit, at which time the procedures normally scheduled for the W16 visit will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥18 years of age.
2. Able and willing to give informed consent and to comply with scheduled visits and trial procedures.
3. A diagnosis of DKD due to either T1DM or T2DM (diagnosed for ≥1 year)
4. On a stable anti-diabetic medication regimen for ≥4 months prior to randomization with a hemoglobin A1C (HbA1c) <9.5%.

   1. Participants with T1DM may not be on any glucose lowering medications beyond insulin.
   2. Participants with T2DM may be on more than 1 anti diabetic medication regimen (eg, SGLT2 inhibitor, insulin, or other anti-diabetic medication regimen).
   3. HbA1c should have been performed within the last 4 months prior to randomization.
5. Participants must be on a stable dose of ACEi or ARB for ≥4 months prior to randomization and expected to remain stable for the 4-month treatment period.
6. Participants taking finerenone (not required), on a stable dose for ≥4 months prior to randomization.
7. Presence of albuminuria with a UACR >100 mg/g and <3000 mg/g at screening.

Exclusion Criteria:

1. Significant medical condition, that in the opinion of the Investigator will place the participant at risk during the study or that will confound the study endpoints.
2. Participants not fully vaccinated for Coronavirus Disease 2019 (COVID 19).

   1. Participants will be considered fully vaccinated if they have received all recommended doses of a COVID-19 vaccine that has been authorized or approved by the United States Food and Drug Administration (FDA) or is listed for emergency use by the World Health Organization within 14 days prior to the first dose of the study drug.
   2. Participants who have fully recovered from COVID 19 and have a negative COVID-19 test ≥14 days before screening are eligible.
3. Other causes of kidney disease that are not DKD (eg, lupus nephritis). Of note, hypertension is not an exclusion criteria.
4. Participants with an eGFR <30 ml/min/1.73m².
5. Participants who have had acute kidney injury (AKI) within the past 3 months, or have ever received dialysis.
6. Participants with a history of epilepsy or intracranial surgery.
7. Uncontrolled hypertension with measurements of systolic pressures >160 or diastolic measurements >100 at the Screening Visit.
8. Active substance abuse including inhaled or injection drugs in the year prior to screening.
9. Use of cannabis or cannabinoid containing compounds within 90 days prior to screening.
10. Pregnancy, planned pregnancy, potential for pregnancy or unwillingness to use effective birth control during the trial, as well as breast feeding.
11. Evidence of moderate to severe hepatic impairment as defined by Child's-Pugh B or C.
12. Subjects with a history of significant psychiatric disorder, including but not limited to:

    1. Major depression within the last 2 years.
    2. Any history of a suicide attempt or suicidal ideation.
    3. Subjects with a history of other severe psychiatric disorders (eg, schizophrenia, bipolar disorder).
13. Score of the 9-question Patient Health Questionnaire (PHQ-9) ≥15 at baseline.
14. Current or active malignancy within the past 5 years, except for cancer in situ, or non-melanoma skin cancer such as basal cell or squamous cell carcinoma that has been completely resected.
15. QTc >500 msec at baseline.
16. Any chronic medications started or changed within the past 3 months or at risk of needing to be changed during the study.
17. Participants with a history of hyperthyroidism or other thyroid diseases.
18. Participants taking a strong inducer or inhibitor of cytochrome P450 3A4, 2D6 or 2C19 by screening. These medications are prohibited during the entire study duration.
19. Having taken any investigational compound within 30 days, or 5 half-lives of the drug, whichever is longer, before the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Change in UACR from baseline to W16 | 16 weeks
  Measure of UACR at W16 in comparison to baseline to evaluate the effect of INV-202 in participants with diabetic kidney disease (DKD)

SECONDARY OUTCOMES:
Change in urine protein to creatinine ratio (UPCR) from baseline to W16 | 16 weeks
  Measure of UPCR at W16 in comparison to baseline to evaluate the effect of INV-202 in participants with diabetic kidney disease (DKD)
Change in eGFR using serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula from baseline to W16 | 16 weeks
  Measure of eGFR using creatinine and CKD-EPI formula at W16 in comparison to baseline to evaluate the effect of INV-202 in participants with diabetic kidney disease (DKD)
Change in eGFR using cystatin C and the CKD-EPI formula from baseline to W16 | 16 weeks
  Measure of eGFR using cystatin C and CKD-EPI formula at W16 in comparison to baseline to evaluate the effect of INV-202 in participants with diabetic kidney disease (DKD)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Crater, MD, Study Director — Inversago Pharma
Locations (70):
- United States (22):
  - National Institute of Clinical Research, Inc., Garden Grove, California
  - National Institute of Clinical Research, Inc - Pomona, Pomona, California
  - Central Coast Nephrology, Salinas, California
  - North American Research Institute, San Dimas, California
  - National Institute of Clinical Research, Inc - Upland, Upland, California
  - Research Physicians Network Alliance, Boca Raton, Florida
  - ALL Medical Research, LLC, Cooper City, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Research by Design, LLC, Chicago, Illinois
  - Endocrine and metabolic Consultants, Rockville, Maryland
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Palm Research Center, Inc, Las Vegas, Nevada
  - Physicians East, PA, Greenville, North Carolina
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - South Carolina Clinical Research LLC, Orangeburg, South Carolina
  - Knoxville Kidney Center, Pllc, Knoxville, Tennessee
  - North Texas Endocrine Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Linq Research, LLC, Pearland, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
- Canada (2):
  - Centre de recherche Clinique de Laval, Laval, Quebec
  - GCP Research, Montreal, Quebec
- Georgia (14):
  - "Clinic- LJ", LTD, Kutaisi
  - LTD Clinic Rustavi, Rustavi
  - L. Managadze National Center of Urology, LTD, Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center LTD, Department of Internal Medicine and Medical Research, Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center LTD, Department of Multi-center Clinical Trials, Tbilisi
  - Archangel St Michael Multiprofile Clinical Hospital Ltd, Tbilisi
  - Ltd "Institute of Clinical Cardiology", Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - Georgian Dutch Hospital LLC, Tbilisi
  - LTD Tbilisi Heart Center, Tbilisi
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - Israel-Georgia Research Clinic Helsicore, LTD, Tbilisi
  - LTD "Adapt", Tbilisi
  - National Institute of Endocrinology, LTD,, Tbilisi
- Hungary (5):
  - Diaverum Dialysis Centre of Baja and Nephrology Out-Patient Clinic of Baja St.Rokus Hospital, Baja
  - DPC Hospital - Central Hospital of Southern Pest National Institute of Hematology and Infectious Diseases, 1st Department of Internal Medicine, Budapest
  - University of Debrecen, Debrecen
  - Flor Ferenc Hospital of Pest County, Kistarcsa
  - Medifarma-98 Kft, Nyíregyháza
- Israel (9):
  - Haemek medical center, Afula
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus \ Rambam Medical Center, Haifa
  - Wolfson medical center, Holon
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Ziv Medical Center - Endocrinology Clinic, Safed
  - Ziv Medical Center, Safed
- Mexico (9):
  - Instituto de Diabetes Obesidad Y Nutricion , S.C., Cuernavaca
  - Centro de Investigación Médica y Reumatología S.C., Guadalajara
  - Cento de Investigacion Medica de Occidente, S.C., Guadalajara
  - Medical Office, Guadalajara
  - Unidad de Investigación Clinica y atencion Medica HEPA, Guadalajara
  - Clinica Integral del Paciente Diabético y Obeso, Mexico City
  - Investigación Médica, Mérida
  - St Lucas Clinical Research Center SA de CV, Mérida
  - Instituto Veracruzano en Investigacion Clínica S.C., Veracruz
- Serbia (9):
  - Clinical Hospital Center Zemun, Belgrade
  - General Hospital "Vršac", Belgrade
  - University Clincial Center of Serbia, Belgrade
  - University of Kragujevac - Klinicki Centar "Kragujevac", Kragujevac
  - General Hospital Krusevac, Kruševac
  - University Clinical Center Nis, Clinic of Nephrology, Niš
  - University Clinical Center of Vojvodina, Novi Sad
  - Healt Center Uzice,General Hospital, Užice
  - Health Center Zajecar, Zaječar

IPD SHARING:
Plan to Share IPD: No